CLINICAL TRIAL: NCT06596551
Title: Aspirational Rehabilitation Coaching for Holistic Health (ARCH): A Pilot Pre-Post Evaluation of Psychosocial Recovery in First-Time Stroke Survivors and Family Caregivers
Brief Title: Aspirational Rehabilitation Coaching for Holistic Health (ARCH): A Pilot Pre-Post Experimental Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Collaborators: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Andy Hau Yan Ho, PhD, EdD, Professor, Nanyang Technological University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2023-00-355
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Psychological Well-Being; Psychosocial Functioning
MeSH Terms: conditions — Stroke; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Pre-post single arm study design will measure psychosocial health outcomes before and again after the intervention is implemented. This study design is adopted for the purposes of a pilot investigation to observe if the ARCH intervention can have temporary effects or no effects on psychosocial health outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-Post ARCH Intervention (Experimental): Participants will receive the ARCH intervention, a 4-weekly, 6-hour, strength-based dyadic programme that integrates psychoeducation, psychosocial support, and self-compassion practices to encourage and inspire families recovering from a first-time stroke. Specific intervention components include family education, facilitated dyadic communication and mindful self-compassion practices. Weekly therapeutic objectives build upon each other to provide affected families with the necessary means to process the trauma of experiencing a stroke and learning to live amidst multiple post-stroke losses.
  Interventions: Behavioral: Pre-Post ARCH Intervention

INTERVENTIONS:
Behavioral: Pre-Post ARCH Intervention — Stroke dyads, consisting of a survivor and primary family caregiver, will engage in a 4 weekly, 1.5 hour experiential dyadic sessions, totalling 6 hours of participation. In Week 1, dyads acknowledge the losses occurring after the stroke to normalize feelings of grief and sadness and find comfort within the familial space. In Week 2, dyads interpret their post-stroke losses within the framework of their existing knowledge for managing adversities (strengths, resources, and values) and identify changes that are most meaningful to them. In Week 3, dyads set specific, measurable, and achievable goals to actualize the meaningful changes identified in Week 2. Finally in Week 4, dyads bring together their individually derived strengths from the previous sessions to culminate into strengthened dyadic bonds. The exercise will also encourage participants to expand beyond the dyadic space to seek support from their communities, social networks and care services that are available to them.

SUMMARY:
The ARCH programme is a novel, strength-based, dyadic, multicomponent psychosocial intervention that blends together psychoeducation, psychosocial support and self-compassion practices to aid first-time stroke survivors and their family caregivers with their psycho-socio-emotional and spiritual challenges following discharge from in-patient care. A pre-post experimental design with a feasibility and acceptability assessment is adopted to evaluate and refine the ARCH intervention in promoting wellbeing, self-compassion, independence, quality of life, hope, resilience, self-efficacy and dyadic mutuality.

DETAILED DESCRIPTION:
Objective: The current study utilizes the empirical foundations of psychosocial recovery in first-time stroke dyads to pilot test the Aspirational Rehabilitation Coaching for holistic Health (ARCH) programme. The core objectives of this study is to 1) critically assess the pre-post effects in participants' psycho-socio-emotional and spiritual wellbeing and 2) qualitatively evaluate the feasibility and acceptability of the intervention in addressing post-stroke psychosocial challenges.

Methods: For this pilot study a total of 30 survivor-caregiver dyads (N=60; 30 survivors, 30 caregivers) will be recruited directly through referrals from the collaborating hospital. The proposed sample size reflects the approximate or working number of qualitative interviews at which one could expect to be reach theoretical saturation (Morse, 2000). Participants above the ages of 21 years, recovering from their first stroke at mild to moderate degree of severity, discharged from inpatient care at no later than 3 months, clinically assessed to have cognitive capacities to engage in and complete the research study, with language capabilities in English or Mandarin and one identified primary family caregiver over the age of 21 will be recruited for this study. Consenting family dyads will undergo a 4-week dyadic intervention that integrates psychoeducation, psychosocial support, and self-compassion practices. The rationale for the intervention components was based on an in-depth analysis of the psychosocial needs and challenges of stroke survivors and family caregivers reported in the international literature, and the lived experiences of post-stroke loss, coping strategies and recovery needs of Singaporean first-time stroke survivors and family caregivers. Quantitative measurements will be taken at baseline [time point 1 (T1)], immediately after the intervention [T2], 3 months [T3] and 6 months [T4] post-intervention. The qualitative assessment of feasibility and acceptability will be conducted at post intervention [T2].

Significance: The absence of tailored, family-centered support in current stroke rehabilitation practices suggest that more and more individuals are left to their own devices in navigating this psychologically, socially, and emotionally devastating health event. Dyads participating in this study will experience, for the first time ever, a rehabilitative programme that is solely focused in providing them the comfort and support in managing their unique psycho-socio-emotional and spiritual challenges post-stroke. Results from this study hope to inform the large stroke community and eventually find advocate for the ARCH intervention to become a part of standard clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years and above
* Recovering from their first stroke at mild to moderate degree of severity
* Discharged from inpatient care at no later than 3 months,
* Clinically assessed to have cognitive capacities to engage in and complete the research study,
* Language capabilities in English or Mandarin, and
* One identified primary family caregiver aged 21 years and above with similar language capabilities.

Exclusion Criteria:

* Families with survivors suffering from aphasia,
* Being too ill to participate,
* Experiencing moderate to severe cognitive impairment, and
* With family caregivers who are not interested to participate.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in well-being from baseline (patient) | Participants will be assessed at four time points: [T1] baseline; [T2] immediately post-intervention; [T3] 3 months post-intervention; and [T4] 6 months post-intervention
  The 7-item short version of the Warwick Edinburgh Mental Well-being Scale (SWEMWBS) is a measure of mental well-being. Participants will be assessed on a 5-point scale.
Change in well-being from baseline (caregiver only) | Participants will be assessed at four time points: [T1] baseline; [T2] immediately post-intervention; [T3] 3 months post-intervention; and [T4] 6 months post-intervention
  The 8-item short version of the WHOQOL-100 and the WHOQOL-BREF, that assesses four domains of quality of life (psychological, physical, social, and environmental). Participants will be assessed on a 5-point scale.
Change in post-stroke reintegration from baseline (patient only) | Participants will be assessed at four time points: [T1] baseline; [T2] immediately post-intervention; [T3] 3 months post-intervention; and [T4] 6 months post-intervention
  The Modified Reintegration to Normal Living Index (mRNLI) is a 11-item questionnaire that evaluates reintegration to normal living after incapacitating illness or trauma on a 4-point scale.
Change in caregiver burden from baseline (caregiver only) | Participants will be assessed at four time points: [T1] baseline; [T2] immediately post-intervention; [T3] 3 months post-intervention; and [T4] 6 months post-intervention
  The Zarit Burden Interview Short (ZBI-Short) is a 12-item questionnaire that assesses caregiver burden on a 4-point scale.
Change in self-efficacy from baseline (patient only) | Participants will be assessed at four time points: [T1] baseline; [T2] immediately post-intervention; [T3] 3 months post-intervention; and [T4] 6 months post-intervention
  The General Self-Efficacy Scale (GSES) is a 10-item questionnaire that utilizes a 4-point scale to measure perceived self-efficacy is areas of goal setting, effort investment, persistence in face of barriers and recovery from setbacks.

SECONDARY OUTCOMES:
Changes in dyadic relationship interactions from baseline | Participants will be assessed at four time points: [T1] baseline; [T2] immediately post-intervention; [T3] 3 months post-intervention; and [T4] 6 months post-intervention
  The Dyadic Relationship Scale (DRS) utilizes a 4-point scale to measure both the patient and the family caregiver's perspectives on the positive and negative aspects of their dyadic interactions.
Change in spiritual well-being from baseline | Participants will be assessed at four time points: [T1] baseline; [T2] immediately post-intervention; [T3] 3 months post-intervention; and [T4] 6 months post-intervention
  The Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being (FACIT-Sp-12) is a 12-item questionnaire that utilizes a 4-point scale to measure overall spiritual well-being and it's components on three sub-scales (faith, meaning and peace).
Change in anxiety and depression symptoms from baseline | Participants will be assessed at four time points: [T1] baseline; [T2] immediately post-intervention; [T3] 3 months post-intervention; and [T4] 6 months post-intervention
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire that utilizes a 4-point scale to measure symptoms of psychological distress in non-psychiatric clinical settings.
Changes in perception of social support from baseline | Participants will be assessed at four time points: [T1] baseline; [T2] immediately post-intervention; [T3] 3 months post-intervention; and [T4] 6 months post-intervention
  The Lubben Social Network Scale 6 (LSNS-6) is a 6-item questionnaire that utilizes a 6-point scale to assess social networks, available social support and screen for social isolation
Change in resilience from baseline | Participants will be assessed at four time points: [T1] baseline; [T2] immediately post-intervention; [T3] 3 months post-intervention; and [T4] 6 months post-intervention
  The Brief Resilience Scale (BRS) is a 6-item questionnaire that utilizes a 5-point scale to assess an individual's perceived ability to bounce back or recover from stress.
Change in hope from baseline | Participants will be assessed at four time points: [T1] baseline; [T2] immediately post-intervention; [T3] 3 months post-intervention; and [T4] 6 months post-intervention
  The Herth Hope Index (HHI) is a 12-item questionnaire that utilizes a 4-point scale to measure hope in clinical settings with terminally ill adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choo PY, Shaik MA, Tan-Ho G, Lee J, Ho AHY. Living losses in stroke caregiving: A qualitative systematic review of systematic reviews on psycho-socio-emotional challenges and coping mechanisms. Int J Stroke. 2023 Mar;18(3):268-277. doi: 10.1177/17474930221104908. Epub 2022 Jul 5. PMID 35619566
- [Background] da Rocha NS, Power MJ, Bushnell DM, Fleck MP. The EUROHIS-QOL 8-item index: comparative psychometric properties to its parent WHOQOL-BREF. Value Health. 2012 May;15(3):449-57. doi: 10.1016/j.jval.2011.11.035. Epub 2012 Feb 9. PMID 22583455
- [Background] Herth K. Abbreviated instrument to measure hope: development and psychometric evaluation. J Adv Nurs. 1992 Oct;17(10):1251-9. doi: 10.1111/j.1365-2648.1992.tb01843.x. PMID 1430629
- [Background] Tang JY, Ho AH, Luo H, Wong GH, Lau BH, Lum TY, Cheung KS. Validating a Cantonese short version of the Zarit Burden Interview (CZBI-Short) for dementia caregivers. Aging Ment Health. 2016 Sep;20(9):996-1001. doi: 10.1080/13607863.2015.1047323. Epub 2015 May 27. PMID 26016419
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Haver A, Akerjordet K, Caputi P, Furunes T, Magee C. Measuring mental well-being: A validation of the Short Warwick-Edinburgh Mental Well-Being Scale in Norwegian and Swedish. Scand J Public Health. 2015 Nov;43(7):721-7. doi: 10.1177/1403494815588862. Epub 2015 Jun 3. PMID 26041133
- [Background] Miller A, Clemson L, Lannin N. Measurement properties of a modified Reintegration to Normal Living Index in a community-dwelling adult rehabilitation population. Disabil Rehabil. 2011;33(21-22):1968-78. doi: 10.3109/09638288.2011.553707. Epub 2011 Feb 9. PMID 21306195
- [Background] Minshall C, Castle DJ, Thompson DR, Pascoe M, Cameron J, McCabe M, Apputhurai P, Knowles SR, Jenkins Z, Ski CF. A psychosocial intervention for stroke survivors and carers: 12-month outcomes of a randomized controlled trial. Top Stroke Rehabil. 2020 Dec;27(8):563-576. doi: 10.1080/10749357.2020.1738677. Epub 2020 Mar 19. PMID 32191569
- [Background] Sebern MD, Whitlatch CJ. Dyadic relationship scale: a measure of the impact of the provision and receipt of family care. Gerontologist. 2007 Dec;47(6):741-51. doi: 10.1093/geront/47.6.741. PMID 18192628
- [Background] Peterman AH, Fitchett G, Brady MJ, Hernandez L, Cella D. Measuring spiritual well-being in people with cancer: the functional assessment of chronic illness therapy--Spiritual Well-being Scale (FACIT-Sp). Ann Behav Med. 2002 Winter;24(1):49-58. doi: 10.1207/S15324796ABM2401_06. PMID 12008794
- [Background] Lubben J, Blozik E, Gillmann G, Iliffe S, von Renteln Kruse W, Beck JC, Stuck AE. Performance of an abbreviated version of the Lubben Social Network Scale among three European community-dwelling older adult populations. Gerontologist. 2006 Aug;46(4):503-13. doi: 10.1093/geront/46.4.503. PMID 16921004
- [Background] Kurimoto A, Awata S, Ohkubo T, Tsubota-Utsugi M, Asayama K, Takahashi K, Suenaga K, Satoh H, Imai Y. [Reliability and validity of the Japanese version of the abbreviated Lubben Social Network Scale]. Nihon Ronen Igakkai Zasshi. 2011;48(2):149-57. doi: 10.3143/geriatrics.48.149. Japanese. PMID 21778631
- [Background] Fung SF. Validity of the Brief Resilience Scale and Brief Resilient Coping Scale in a Chinese Sample. Int J Environ Res Public Health. 2020 Feb 16;17(4):1265. doi: 10.3390/ijerph17041265. PMID 32079115